CLINICAL TRIAL: NCT03166488
Title: Evaluation of Liver Stiffness After Tricuspid Valvular Repair Using Magnetic Resonance Elastography
Brief Title: MRE Evaluation of Liver Stiffness After Tricuspid Valvular Repair
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael L Wells, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-009548
Record Dates: First submitted 2017-05-19; First posted 2017-05-25 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Tricuspid Valve Insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Tricuspid Valvular Repair Patients (Experimental): Subjects will receive an MRI sequence called Magnetic Resonance Elastography (MRE) within 1 month preoperatively and as close to 6 months postoperatively as reasonably achievable.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Subjects will receive an MRI sequence called Magnetic Resonance Elastography (MRE).

SUMMARY:
The purpose of this study is to look at liver stiffness with a MRI sequence called Magnetic Resonance Elastography (MRE). The study will let the investigators know whether the subject's liver is normal or has increased stiffness. Increased liver stiffness often means there is chronic liver disease and fibrosis. Increased right heart pressure and congestive heart failure are considered risk factors for development of liver fibrosis. Liver fibrosis, if progressive, may lead to cirrhosis and its related complications. The increased liver stiffness may be due to a poorly functioning tricuspid valve. With this research, the investigators will be able to determine if the elevated stiffness of the liver returns to normal after the surgeon performs a repair or replacement of the tricuspid valve.

ELIGIBILITY:
Inclusion criteria:

* Primary tricuspid valvular regurgitation (tricuspid valve disease not related to a left-sided cardiac abnormality) diagnosed by echocardiography
* Evidence of passive hepatic congestion. Patients with severe tricuspid regurgitation diagnosed at echocardiography will constitute evidence of passive hepatic congestion.
* Patient scheduled for surgical tricuspid valvular repair or replacement.

Exclusion criteria:

* Contraindication for MRI (implantable devices such as cardiac pacemaker, anxiety, inability to lay supine, etc).
* Additional conditions which may elevate their liver stiffness: hepatic fibrosis or cirrhosis, hepatic parenchymal disease (primary biliary cirrhosis, primary sclerosing cholangitis, etc), acute or chronic hepatitis (viral, substance or medication induced), disorders of hepatic vasculature, biliary obstruction or disease, primary or metastatic hepatic malignancy.
* Cannot agree to return for a follow up visit to complete the postsurgical imaging.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in liver stiffness between preoperative and postoperative MR elastography (MRE) | baseline, approximately 6 months postoperatively
  Increased liver stiffness often means there is chronic liver disease and fibrosis.
Change in tricuspid valve regurgitation measured by echocardiography | baseline, approximately 6 months postoperatively
  Increased liver stiffness may be due to a poorly functioning tricuspid valve.

SECONDARY OUTCOMES:
Change in Subject Functional Capacity | baseline, approximately 6 months postoperatively
  Subject Functional Capacity will be measured by the Self Assessment New York Heart Association (NYHA) Classification Scale. This questionnaire consists of 4 questions regarding the subject's ability to carry on physical activities. NYHA Class I = no symptoms in regular activity; NYHA Class II = Mild symptoms and slight limitation; NYHA Class III = noticeable limitations even during minimal activity; NYHA Class IV = severe limitations even while at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Wells, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: Undecided